CLINICAL TRIAL: NCT07137715
Title: Pain Reprocessing Therapy for Veterans With Chronic Back Pain: Comparative Efficacy and Facilitators and Barriers to Implementation
Brief Title: Psychological Options for Wellness and Recovery (POWeR) Trial for Veterans With Chronic Back/Neck Pain
Acronym: POWeR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: VA Eastern Colorado Health Care System (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-2398; HT9425-24-1-0915 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-08-11; First posted 2025-08-22 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Chronic Pain; Back Pain; Back Pain Lower Back Chronic; Neck Pain
Keywords: Pain Reprocessing Therapy (PRT); PRT; Chronic Pain; Veterans; Neck Pain; Back Pain; Cognitive Behavioral Therapy (CBT); CBT
MeSH Terms: conditions — Chronic Pain; Back Pain; Neck Pain | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: Three-arm randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessment will be completed via automated transmission of a REDCap link, and as such is inherently blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pain reprocessing therapy (PRT) (Experimental): PRT has 5 components: 1) education about the origin of pain in the brain, its reversibility, and the pain-fear cycle; 2) reinforcing education using personal biography; 3) "somatic tracking" of pain through mindfulness and reappraisal of pain sensations as non-dangerous; 4) lowering the level of personal threat that may trigger pain sensation; and 5) inducing positive affect in periods of pain. Patients will attend 1 assessment and education telehealth session with a physician followed by 8, 50-minute, therapist-led sessions. Pacing will be weekly for approximately 9 weeks. Treatment will be provided by experienced PRT clinicians. All PRT sessions will be remotely-delivered.
  Interventions: Behavioral: Pain reprocessing therapy (PRT)
- Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) (Active Comparator): CBT-CP, considered the leading psychological treatment for chronic pain, is a structured, time-limited intervention that aims to teach patients how to better manage chronic pain and improve their quality of life. Participants will receive 9, 50-minute sessions of CBT-CP over 9 weeks. The VA CBT-CP protocol contains an initial orientation involving education and familiarization with the CBT-CP approach to chronic pain. The protocol then includes sessions that focus on topics such as exercise, relaxation, pleasant activities, cognitive coping, and sleep. All CBT-CP sessions will be remotely-delivered.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Chronic Pain (CBT-CP)
- Usual Care (Active Comparator): Participants will be asked to continue whatever they are already doing to care for their back pain. Length of the usual care condition will be 9 weeks, the expected completion time of the PRT and CBT arms.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Pain reprocessing therapy (PRT) — A promising new psychotherapy for chronic pain
  Arms: Pain reprocessing therapy (PRT)
Behavioral: Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) — A psychotherapy for chronic pain that has 30+ years of research support.
  Other Names: Cognitive Behavioral Therapy (CBT)
  Arms: Cognitive Behavioral Therapy for Chronic Pain (CBT-CP)
Other: Usual Care — Participants will be asked to continue to do whatever they are currently doing to manage their pain.
  Other Names: Treatment as usual
  Arms: Usual Care

SUMMARY:
The goal of this clinical trial is to learn which treatment works better for veterans with chronic neck or back pain. This study is comparing three treatments: Pain Reprocessing Therapy (PRT), Cognitive Behavioral Therapy (CBT), and usual care (whatever a person is already doing to cope with their pain).

The main questions the study aims to answer are:

1. Which treatment works better for lowering pain: PRT, CBT, or usual care?
2. How do the effects of PRT compare with CBT and usual care in terms of pain relief and other factors such as emotional functioning, quality of life, anxiety, and pain medication use?

Participants will:

1. Be randomly assigned to receive either PRT, CBT, or usual care.
2. Complete questionnaires about their pain and health.
3. If in the PRT or CBT group, have nine weekly therapy sessions over video calls with a therapist.

DETAILED DESCRIPTION:
The current leading psychotherapeutic treatment for chronic pain is cognitive behavioral therapy (CBT-CP), which has been found to be safe and modestly efficacious in the treatment of chronic back or neck pain (CBNP). The fundamental goal of CBT-CP is to encourage participants to adopt an active, problem-solving approach to managing the challenges associated with chronic pain. CBT-CP intervention follows a standard structure of 9 sessions with the following objectives: 1) reducing the negative impact of pain on daily life 2) improving physical and emotional functioning 3) increasing effective coping skills for managing pain 4) reducing pain intensity. Recent evidence shows CBT provides a 1-1.5 point reduction in pain intensity on an 11-point pain scale when compared to treatment as usual.

Using advances in neuroscience and psychology, investigators recently developed a novel psychological treatment called Pain Reprocessing Therapy (PRT). Using a combination of cognitive, exposure-based, and somatic psychotherapy techniques, PRT aims to promote patients' reconceptualization of pain as due to reversible, non-dangerous brain activity rather than peripheral pathology. Critically, PRT aims to reduce or eliminate pain, rather than merely increase functioning.

In the first trial of PRT (N = 151), 66% of patients randomized to PRT were pain-free or nearly pain-free at post-treatment, compared to fewer than 20% of those in the placebo and usual care control groups. PRT has several critical conceptual distinctions from CBT including different approaches to pain subtyping, a different understanding of chronic pain etiology, differing treatment goals (recovery vs. improved functioning), and a different focus on non-pain psychosocial threats. Given the conceptual differences and early existing promising efficacy data of PRT, a critical next step to achieve practical improvements in Veteran health is a comparative effectiveness trial of PRT vs. CBT in a Veteran Affairs (VA) clinic, utilizing VA clinicians, VA treatment infrastructure, and Veteran participants.

Aim 1 of this study is to test the comparative effectiveness of PRT to CBT and usual care on pain severity (primary outcome) for veterans with CBNP at post-treatment (primary endpoint) and one year follow-up.

Aim 2 of this study is to test the comparative effectiveness of PRT to CBT and usual care on secondary patient-reported outcomes measuring core outcome domains, quality of life, and opioid medication use.

Aim 3 of this study is to identify key barriers and facilitators of PRT response in a Veteran population using qualitative methods in a subsample of participants (n = 40) and in clinicians learning PRT.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 and older)
* Be veterans
* Have a history of chronic back or neck pain defined as pain at least half the days of the last 6 months.
* Have moderate or greater pain, defined as pain intensity ≥4 in the past week

Exclusion Criteria:

Clinical presentation suggestive of back pain that is secondary or peripheral in nature, including self-reported leg pain that is worse than back pain (indicative of radiculopathy or sciatica), spine surgery within the past 6 months, fall, motor vehicle accident or other trauma related to back pain in the past 6 months, back pain due to an inflammatory disorder, infection, or malignant etiology as determined per medical provider review, known sensory abnormality in trunk or legs, recent large (>20 lbs) unexplained weight loss, difficulty controlling bowels (to screen out cauda equina syndrome), and self-reported diagnoses of specific inflammatory disorders (rheumatoid arthritis, polymyalgia rheumatica, scleroderma, Lupus, and polymyositis).

Additionally, patients who meet any of the following criteria are ineligible due to anticipated difficulties complying with study procedures:

* Moderate or severe cognitive impairment
* Unstable or severe untreated mental health condition, including active suicidal ideation
* Unstable or end-stage medical disease including active cancer
* Back surgery planned within the next 6 months
* Inability to communicate by telephone or video, including inability due to housing instability
* Current pain-related litigation outside the VA (service connection-related applications are not excluded)
* Having engaged in CBT or PRT for chronic pain in the past 6 months
* Participants may be excluded based on the discretion of PIs Ashar and Frank

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Post-treatment (at an average of 10 weeks) and 26, 39, and 52 weeks post-randomization
  Last-week average pain intensity is assessed via the Brief Pain Inventory Short Form (BPI-SF). The BPI-SF assesses pain severity and its impact on functioning. It consists of 9 total items including 4 pain intensity items and 5 pain interference items. The 4 pain intensity items measure pain in the last week on a numerical rating scale of 0 (no pain at all) to 10 (pain as bad as you can imagine).

SECONDARY OUTCOMES:
Pain Interference | Post-treatment (at an average of 10 weeks) and 26, 39, and 52 weeks post-randomization
  Last-week average pain interference is assessed via the Brief Pain Inventory Short Form (BPI-SF). The BPI-SF assesses pain severity and its impact on functioning. It consists of 9 total items including 4 pain intensity items and 5 pain interference items. The 5 pain interference items measure the impact of pain on General Activity, Mood, Walking Ability, Normal Work, Relations with other people, Sleep, and Enjoyment of Life. Each area is rated on a numerical rating scale from 0 (does not interfere) to 10 (completely interferes).
Satisfaction with Life | Post-treatment (at an average of 10 weeks) and 26, 39, and 52 weeks post-randomization
  Satisfaction with Life is assessed via the self-reported 5-Item Satisfaction with Life Scale (SWLS). The SWLS measures an individual's global life satisfaction. Each item is rated on a 7-point Likert scale (1=Strongly Disagree and 7=Strongly Agree). The ratings are summed to determine an overall score.
Depression | Post-treatment (at an average of 10 weeks) and 26, 39, and 52 weeks post-randomization
  Depression is assessed using the self-reported 4-item Patient-Reported Outcomes Measurement Information System Depression Short Form 4a (PROMIS-Depression-SF 4a). The individual items measure negative mood, loss of interest, helplessness, and hopelessness over the past 7 days. Each item is scored 1-5, and raw scores are then converted to a T-score using pre-determined cut-offs.
Anxiety | Post-treatment (at an average of 10 weeks) and 26, 39, and 52 weeks post-randomization
  Anxiety is assessed using the self-reported 4-item Patient-Reported Outcomes Measurement Information System Anxiety Short Form 4a (PROMIS-Anxiety-SF 4a). The form's items measure an individual's fear, worry, tension, and difficulty concentrating over the past 7 days. Each item is scored 1-5, and raw scores are then converted to a T-score using pre-determined cut-offs.
Fatigue | Post-treatment (at an average of 10 weeks) and 26, 39, and 52 weeks post-randomization
  Fatigue is assessed using the self-reported 4-item Patient-Reported Outcomes Measurement Information System Fatigue Short Form 4a (PROMIS-Fatigue-SF 4a). The form's items measure an individual's fatigue intensity, fatigue frequency, fatigue-related difficulty initiating actions, and feelings of energy depletion. Each item is scored 1-5, and raw scores are then converted to a T-score using pre-determined cut-offs.
Post-Traumatic Stress Disorder (PTSD) Symptoms | Post-treatment (at an average of 10 weeks) and 26, 39, and 52 weeks post-randomization
  PTSD symptoms are assessed using the self-reported 6-item Primary Care PTSD Screen for DSM-5 (PC-PTSD-5). All items are Yes/No questions. The first item screens whether the respondent has experienced a traumatic event, and the other five items assess how this trauma has affected them over the past month. The score is the number of Yes answers to the last five items. Respondents who answer No to the first item receive a score of 0 and do not answer the remaining items.
Client satisfaction | Post-treatment (at an average of 10 weeks) and 26, 39, and 52 weeks post-randomization
  Client Satisfaction is assessed the Patients' Global Impression of Change (PGIC). The PGIC is a three-item self-report scale that measures a patient's belief about the efficacy of treatment for their physical health, emotional health, and pain severity. Each item is rated on a 7-point scale of 1 (Very much worse) to 7 (Very much improved).
Medication Use | Post-treatment (at an average of 10 weeks) and 26, 39, and 52 weeks post-randomization
  Medication use is assessed in two ways: 1) electronic health record review and 2) patient self-report of past-week frequency of medication, drug, or supplement use to manage pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan K. Ashar, PhD, Principal Investigator — University of Colorado, Denver; Joseph W. Frank, MD, MPH, Principal Investigator — VA Eastern Colorado Health Care System
Locations (1):
- VA Eastern Colorado Health Care System, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing procedures have not been finalized. At a minimum, a complete, cleaned, de-identified copy of the final dataset used in conducting the final analyses of the study will be created and made available within one year after the completion of the study, pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset. Depending on feasibility and guidance from VA Office of Research Oversight, a Limited Dataset (LDS) may be created and shared. We have not yet determined how to operationalize data sharing for this study. In the interim, contact the PI for questions or requests.
Supporting Information: Study Protocol, SAP, ICF